CLINICAL TRIAL: NCT00152191
Title: A Randomized Controlled Study of Postoperative Adjuvant Therapy of UFT Compared With CMF in High-risk Women With Axillary Node-negative Breast Cancer (NSAS-BC)
Brief Title: A Randomized Controlled Study of Postoperative Adjuvant Therapy of Uracil-tegafur (UFT) Compared With Cyclophosphamide/Methotrexate/5-fluorouracil (CMF) in Breast Cancer (NSAS-BC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01023001
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tegafur; Uracil; Cyclophosphamide; Methotrexate; Fluorouracil

ARMS (2):
- 1 (Experimental): UFT (uracil, tegafur)
  Interventions: Drug: UFT (uracil, tegafur)
- 2 (Active Comparator): CMF(cyclophosphamide, methotrexate, and fluorouracil)
  Interventions: Drug: cyclophosphamide, methotrexate, and fluorouracil

INTERVENTIONS:
Drug: UFT (uracil, tegafur) — uracil, tegafur was orally administered by 300 mg per square meter per day for 2 years
  Arms: 1
Drug: cyclophosphamide, methotrexate, and fluorouracil — cyclophosphamide:100 mg, po, day 1-14 methotrexate:40 mg/m2, day 1, 8 q28 days x 6 cycles fluorouracil:500 mg/m2, day 1, 8
  Arms: 2

SUMMARY:
This is a randomized controlled study designed to evaluate the relapse-free survival of the UFT group compared with the CMF group. Patients will be randomly assigned to receive either CMF or UFT within 12 weeks after curative resection. To evaluate treatment efficacy, data on recurrence, and survival will be collected for up to 10 years after enrollment of the final patient. To assess safety, data on adverse events will be collected for 2 years after the start of treatment. Patients'quality of life will be assessed by means of a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Performance status 0 or 1 (ECOG)
* Hematopoietic WBC ≥ 4,000/mm^3 Platelet ≥ 100,000/mm^3
* Hepatic AST and ALT ≤ 2.5 times upper limit of normal(ULN) Total bilirubin ≤ ULN
* Renal Creatinine ≤ ULN

Exclusion Criteria:

* Prior anticancer treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 1996-10; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Overall survival, adverse events, and the quality of life | any time

CONTACTS AND LOCATIONS:
Overall Officials: Toru Watanabe, MD, Principal Investigator — Hamamatsu Oncology Center
Locations (1):
- National Cancer Center, 5-1-1, Tsukiji, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Result] Watanabe T, Sano M, Takashima S, Kitaya T, Tokuda Y, Yoshimoto M, Kohno N, Nakagami K, Iwata H, Shimozuma K, Sonoo H, Tsuda H, Sakamoto G, Ohashi Y. Oral uracil and tegafur compared with classic cyclophosphamide, methotrexate, fluorouracil as postoperative chemotherapy in patients with node-negative, high-risk breast cancer: National Surgical Adjuvant Study for Breast Cancer 01 Trial. J Clin Oncol. 2009 Mar 20;27(9):1368-74. doi: 10.1200/JCO.2008.18.3939. Epub 2009 Feb 9. PMID 19204202